CLINICAL TRIAL: NCT04958174
Title: A Smartphone Application for Screening of Developmental Disorders in Children: a Prospective Feasibility Study
Brief Title: A Smartphone Application for Screening of Developmental Disorders in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Collaborators: Kelindi (Industry)
Responsible Party: Sponsor
Other Study IDs: WP-2021-02
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-06

CONDITIONS: Development, Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users: Users of the web-application
  Interventions: Device: web-application

INTERVENTIONS:
Device: web-application — web application for monitoring children's development
  Other Names: MALO

SUMMARY:
The detection of developmental disorders in the child is often late because the parents do not have the information necessary to consult at the first clinical signs. For example, the diagnosis of autism spectrum disorders is made at the age of 5, so earlier diagnoses are possible earlier or even in the 1st year with appropriate questionnaires.

An application (Malo) has been developed to allow through regular questionnaires from 1 month to 3 years old to assess the child's development by his parents in the form of a digital health record assessing several areas at regular intervals (monthly the 1st year then every 3 to 12 months): sensory, psychomotor development, sleep, height and weight, cognitive and addictions (especially to screens). The questions will be adapted to the age of the child. An alert suggesting to consult the general practitioner or the pediatrician will be generated according to an algorithm validated by a committee of experts.

Based on a study model on health data already carried out as part of the triage application for patients suspected of COVID 19 coronavirus disease.fr with 14 million users in 6 months having improved the relevance of calls to the 15 (8 times fewer unnecessary calls) and general practitioners.

This study will assess parental interest in this application.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child or more under 3 years of age (1 month to 3 years)

Exclusion Criteria:

* Parent of a child who has already been diagnosed with a developmental disorder, known physical or mental disability

Ages: 1 Month to 3 Years | Sex: All
Age Groups: Child
Study Population: The application will be made available to Sarthois after a launch campaign by local media for parents with children aged 1 month to 3 years. The population will include the first 180 users of the application who did not object to the use of their data for this assessment.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
usefulness | 6 months
  number of users who find the application useful

SECONDARY OUTCOMES:
Alert | 6 months
  Description of alerts triggered by algorithms
Consultation | 6 months
  Number of relevant consultations (or teleconsultations) after an alert
postpartum depression | 6 months
  Number of women in postpartum depression

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice DENIS, Pr, Study Director — Weprom
Locations (1):
- ILC, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denis F, Maurier L, Carillo K, Ologeanu-Taddei R, Septans AL, Gepner A, Le Goff F, Desbois M, Demurger B, Silber D, Zeitoun JD, Assuied GP, Bonnot O. Early Detection of Neurodevelopmental Disorders of Toddlers and Postnatal Depression by Mobile Health App: Observational Cross-sectional Study. JMIR Mhealth Uhealth. 2022 May 16;10(5):e38181. doi: 10.2196/38181. PMID 35576565